CLINICAL TRIAL: NCT07137338
Title: A Phase 1 Dose Escalation Trial Evaluating an Intravenously Administered Recombinant Adeno-associated Virus Serotype rh.74 (AAVrh.74) Vector Containing the Human BCL2-associated Athanogene 3 (BAG3) Gene Coding Sequence (RP-A701) in Subjects With Dilated Cardiomyopathy Arising From Pathogenic BAG3 Variants (BAG3-DCM)
Brief Title: A Phase 1 AAV Gene Therapy Trial Evaluating Safety and Preliminary Efficacy of RP-A701 in Subjects With BAG3 Dilated Cardiomyopathy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP-A701-0125
Record Dates: First submitted 2025-07-25; First posted 2025-08-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Dilated Cardiomyopathy (DCM)
Keywords: Cardiomyopathy; Dilated; BAG3 Protein; human; dilated cardiomyopathy; DCM; BAG3; BCL2-associated Athanogene 3; Genetic Cardiomyopathy; Gene Therapy; Heart Failure; Ventricular Arrhythmia; Cardiovascular Diseases; Cardiomyopathies; Heart Diseases; Inherited heart disease; AAVrh.74
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies; Dilatation, Pathologic; Heart Failure; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Intervention Model Description: The single-group study will be composed of up to two sequential dose cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single ascending dose of RP-A701 in up to 2 consecutive cohorts (Experimental): Participants will receive a single intravenous dose of RP-A701 on Day 0 and will be followed for up to two years
  Interventions: Genetic: RP-A701 is a recombinant viral vector composed of an AAV serotype rh.74 (AAVrh.74) capsid encapsulating the transgene, BCL2-associated Athanogene 3 (BAG3)

INTERVENTIONS:
Genetic: RP-A701 is a recombinant viral vector composed of an AAV serotype rh.74 (AAVrh.74) capsid encapsulating the transgene, BCL2-associated Athanogene 3 (BAG3) — One-time treatment with a single ascending dose

SUMMARY:
This is a Phase 1, open-label, dose-escalation trial to characterize the safety, tolerability, and preliminary efficacy of RP-A701 following a single IV administration in high-risk adult patients with BAG3-DCM.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion into the study only if all the following criteria apply:

1. Male or female between 18 and 65 years of age at the time of signing the informed consent
2. Capable of and willing to provide signed informed consent
3. Clinical diagnosis of DCM defined as and requiring each of the following:

   1. Mild to moderate systolic dysfunction (LVEF ≥ 25% and ≤ 45%) by echocardiography or CMR performed within 3 months of enrollment.
   2. Absence of severe coronary artery disease (>70% stenosis) or active myocardial ischemia as the etiology of LV systolic dysfunction
   3. Absence of uncontrolled hypertension, significant cardiac valve disease (i.e., greater than moderate in severity), infiltrative disorder, or systemic disease known to cause cardiomyopathy.
4. Documentation of a pathogenic or likely pathogenic variant in BAG3
5. History of ICD implantation ≥ 3 months prior to enrollment
6. NYHA Class II or III HF symptoms with stable HF therapeutic guideline-directed medical regimen for 30 days prior to enrollment

Exclusion Criteria:

1. CV disease that may be related to a genetic etiology other than a BAG3 pathogenic or likely pathogenic variant.
2. Previous participation in a study of gene transfer or gene editing.
3. I.V. inotropic, vasodilator, or diuretic therapy ≤ 30 days prior to enrollment.
4. History of intracardiac thrombosis or arterial thromboembolic events
5. Severe RV dysfunction assessed by echocardiogram or CMR ≤ 12 months prior to screening
6. LVEF < 25% by echocardiogram or CMR at ≤ 3 months prior to screening
7. NYHA Class I or IV HF

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAE) | Baseline up to End of Study (up to 24 months post-infusion)
  Number of participants with Adverse Events following a single IV dose of RP-A701
Incidence of Treatment-emergent Serious Adverse Events (SAE). | Baseline up to End of Study (up to 24 months post-infusion)
  Number of participants with Serious Adverse Events (SAE) following a single IV dose of RP-A701
Incidence of Dose Limiting Toxicities (DLT). | Baseline up to End of Study (up to 24 months post-infusion)
  Number of participants with Dose Limiting Toxicities (DLT) following a single IV dose of RP-A701

SECONDARY OUTCOMES:
To assess the impact of RP-A701 on features of cardiovascular function. | Baseline up to End of Study (up to 24 months post-infusion)
  Change in measures of LV systolic function, including LV ejection fraction (LVEF), LV global longitudinal strain.
To assess the impact of RP-A701 on features of cardiovascular function. | Baseline up to End of Study (up to 24 months post-infusion)
  Change in peak oxygen consumption (VO2) or ventilatory efficiency (VE/VCO2 slope) by cardiopulmonary exercise test (CPET)
To assess the impact of RP-A701 on features of cardiovascular function. | Baseline up to End of Study (up to 24 months post-infusion)
  Change in 6-minute walk distance.
To assess the extent of RP-A701 transduction and protein expression. | Baseline up to End of Study (up to 24 months post-infusion)
  Change in BAG3 myocardial protein expression
To assess the impact of RP-A701 on features of heart failure (HF). | Baseline up to End of Study (up to 24 months post-infusion)
  Change in symptoms of HF assessed by New York Heart Association (NYHA) class.
To assess the impact of RP-A701 on quality of life. | Baseline up to End of Study (up to 24 months post-infusion)
  Change in Kansas City Cardiomyopathy Questionnaire (KCCQ-12) Overall Summary Score.

IPD SHARING:
Plan to Share IPD: No